CLINICAL TRIAL: NCT05619783
Title: A Phase IIIb, Open Label Extension Study Evaluating The Safety And Tolerability of AMX0035 Up To 108 Weeks In Adult Participants With Amyotrophic Lateral Sclerosis (ALS) Previously Enrolled In Study A35-004 (PHOENIX)
Brief Title: Extension Study Evaluating The Safety And Tolerability of AMX0035
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A35-011
Record Dates: First submitted 2022-10-27; First posted 2022-11-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — sodium phenylbutyrate and taurursodiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): All participants will be treated with oral (or feeding tube) AMX0035 (a fixed-dose combination of Sodium Phenylbutyrate (PB) and taurursodiol). All participants will take 2 sachets daily (one morning dose and one evening dose) starting on Day 1, for the duration of the study (if twice a day dosing is poorly tolerated, dosing interruptions and reductions are further discussed in section 6.3) AMX0035 will be supplied by Amylyx as a carton box containing approximately 1 month supply of single use sachets. Each AMX0035 sachet contains active ingredients in a powder formulation with 3 g PB and 1 g taurursodiol. AMX0035 powder is mixed with water and taken orally (or via feeding tube).
  Interventions: Drug: AMX0035

INTERVENTIONS:
Drug: AMX0035 — Combination of 3 g phenylbutyrate and 1 g taurursodiol
  Other Names: RELYVRIO

SUMMARY:
The primary objective is to evaluate the safety and tolerability of AMX0035 over 108 weeks of open label treatment for participants previously enrolled in Study A35-004 (PHOENIX).

DETAILED DESCRIPTION:
All participants will receive open-label treatment with AMX0035, starting on Day 1 with twice a day oral dosing (once in the morning and once in the evening) for the duration of the study. After the Baseline Visit (Day 1), enrolled participants will complete visits approximately every 12 weeks (± 2 weeks), until Week 108 or the end of treatment (EOT) visit, followed by a safety follow-up approximately 28 days after the last dose. A survival follow-up assessment will be completed every 12 weeks following the EOT visit until time of death or end of study (EOS).

ELIGIBILITY:
Inclusion Criteria:

1. Previous participation in Study A35-004 (PHOENIX), including completion of the randomized controlled phase through Week 48 (this timepoint may be upcoming at the time of screening). Participants who do not complete randomized-controlled phase through Week 48 for medical reasons may be included on a case-by-case basis, in consultation with the Sponsor;
2. Capable of providing informed consent;
3. Capable and willing to follow trial procedures including visits to the trial clinic, remote visits, and survival status reporting requirements;
4. Women of childbearing potential (WOCBP; e.g., not post-menopausal for at least one year or surgically sterile must agree to use adequate birth control for the duration of the trial and 3 months after the last dose of AMX0035;

   1. 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle-stimulating hormone (FSH) levels > 40 mIU/ml (milli-international units per milliliter) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
   2. Acceptable contraception methods for use in this trial are:

      * Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants;
      * Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm);
      * Intrauterine device (IUD);
      * Abstinence (no heterosexual sex);
      * Unique partner who is surgically sterile (men) or not of childbearing potential (female).
5. Women must not be pregnant or planning to become pregnant for the duration of the trial and 3 months after last dose of AMX0035;
6. Men must agree to practice contraception for the duration of the trial and for at least 3 months after last dose of AMX0035;
7. Men must not plan to father a child or to provide sperm for donation for the duration of the trial and 3 months after the last dose of AMX0035

Exclusion Criteria:

1. History of known allergy to phenyl butyrate or bile salts;
2. Abnormal liver function defined as bilirubin levels and/or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 5 times the upper limit of the normal (obtained within 12 weeks from first dose);
3. Renal insufficiency as defined by estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 normal (obtained within 12 weeks from first dose);
4. Pregnant women or women currently breastfeeding;
5. Current severe biliary disease which may result in the Investigator medical judgement in biliary obstruction including for example active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gangrene of the gallbladder, abscess of the gallbladder;
6. History of Class III/IV heart failure (per New York Heart Association - NYHA);
7. Participant under severe salt restriction where the added salt intake due to treatment would put the participant at risk, in the Investigator clinical judgment;
8. Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed consent, according to Investigator judgment;
9. Clinically significant unstable medical condition (other than ALS) (e.g., cardiovascular instability, systemic infection, untreated thyroid dysfunction, severe laboratory test anomaly or clinically significant electrocardiogram [ECG] changes) that would pose a risk to the participant if he/she were to participate in the trial, according to Investigator judgment;
10. Currently enrolled in another trial (excluding Study A35-004 (PHOENIX)) involving use of an investigational therapy (or within 5 plasma half-lives) prior to first dose at Baseline Visit;
11. Implantation of Diaphragm Pacing System (DPS);
12. Currently or previously treated within the last 30 days (or 5 half-lives, whichever is longer) from first dose at the Baseline Visit or planned exposure during the treatment period to any prohibited medications listed in Section 6.7 of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
To assess the Incidence of Treatment-Emergent Adverse Events during treatment with AMX0035 | 108 weeks
  Incidence of all adverse events (AE)s; AEs leading to treatment discontinuation or study withdrawal, and all serious adverse events (SAE)s in participants treated with AMX0035

SECONDARY OUTCOMES:
To assess the impact of long-term treatment with AMX0035 on survival | 108 weeks
  1. Overall survival of all-cause mortality
  2. Ventilation free survival (defined as death, tracheostomy for respiratory distress or permanent non-invasive ventilation [>22 hours per day for 7 consecutive days])

CONTACTS AND LOCATIONS:
Overall Officials: Lahar Mehta, MD, Study Director — Head, Global Clinical Development
Locations (46):
- University Hospitals Leuven, Leuven, Belgium
- France (10):
  - Hospices Civils de Lyon Hôpital Neurologique Pierre Wertheimer Cellule Mutualisée de Recherche Clinique (CMRC), Bron
  - Hopital Gabriel Montpied Service de Neurologie, Clermont-Ferrand
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - CHU de Montpellier, Montpellier
  - Gui de Chauliac, Montpellier
  - CHU Nice, Nice
  - Hôpital de la Salpêtrière, Paris
  - Le Centre Hospitalier Régional Universitaire de Tours, Tours
- Germany (6):
  - Uniklinikum Dresden, Dresden
  - Hannover Medical School, Hanover
  - Jena University Hospital, Jena
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - University Medical Center Rostock, Rostock
  - Ulm University Medical Centre, Ulm
- Trinity College Dublin/Beaumont Hospital, Dublin, Ireland
- Italy (10):
  - Università degli Studi di Bari Aldo Moro, Bari
  - Centro Clinico NEMO, Milan
  - IRCCS - Ospedale San Raffaele, Milan
  - University of Milan Medical School, Milan
  - IRCCS - Istituto Auxologico italiano, Milan
  - Azienda Ospedaliero Universitaria Di Modena, Modena
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - University of Padua, Padua
  - Università degli Studi di Bari Aldo Moro, Tricase
  - University of Torino, Turin
- University Medical Center Utrecht, Utrecht, Netherlands
- Poland (2):
  - Centrum Medyczne Linden, Krakow
  - City Clinic Warsaw, Warsaw
- Centro Hospitalar Universitário Lisboa-Norte, Lisbon, Portugal
- Spain (6):
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge-IDIBELL, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital San Rafael, Madrid
  - Biodonostia Health Research Institute; Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario y Politécnico La Fe, Valencia
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Umeå University Hospital, Umeå
- United Kingdom (6):
  - The Walton Centre NHS Trust, Liverpool
  - King's College London, London
  - UCL Queen Square Institute of Neurology, London
  - University of Plymouth, Plymouth
  - Salford Royal Hospital Barnes Clinical Research Team, Salford
  - Sheffield Institute for Translational Neuroscience (SITraN), Sheffield